CLINICAL TRIAL: NCT04550377
Title: Cannabidiol for Treating PTSD Symptoms and Neurocognitive Impairment in PTSD and PTSD Comorbid With TBI: A Placebo-controlled RCT With Neural-circuit Centered Precision Medicine Prediction of Response.
Brief Title: Cannabidiol as a Treatment for PTSD and PTSD Comorbid With TBI
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: Brockman Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 19-00962
Record Dates: First submitted 2020-07-21; First posted 2020-09-16 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Post Traumatic Stress Disorder; Traumatic Brain Injury
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Brain Injuries, Traumatic | interventions — Cannabidiol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cannabidiol Group 1 (Active Comparator): 40 participants will be titrated to a maximum dose of oral cannabidiol 800 mg daily over 2 weeks for a total of 8 weeks treatment.
  Interventions: Drug: Cannabidiol
- Cannabidiol Group 2 (Active Comparator): 40 participants will be titrated to a maximum dose of oral cannabidiol 400 mg daily over 2 weeks for a total of 8 weeks treatment.
  Interventions: Drug: Cannabidiol
- Placebo Group (Placebo Comparator): 40 participants will be given a placebo for a total of 8 weeks treatment.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cannabidiol — The drug product to be used in this study is an oral formulation of CBD
  Other Names: NANTHEIA™; A1002N5S
  Arms: Cannabidiol Group 1; Cannabidiol Group 2
Drug: Placebo — non-active medication
  Arms: Placebo Group

SUMMARY:
This will be a randomized placebo controlled study to test the efficacy of cannabidiol (CBD) as a treatment for symptoms of post-traumatic stress disorder (PTSD). Subjects, 120 in total, will be males and females with PTSD, half of which will have comorbid mild traumatic brain injury (TBI). There will be three study arms, each with 40 subjects: 1) Oral CBD 400 mg daily; 2) Oral CBD 800 mg daily, and 3) Placebo daily. Treatment duration will be 8 weeks. The primary outcome will be change in PTSD symptoms as measured by change in the Clinician-Administered PTSD Scale (CAPS-5) total score.

ELIGIBILITY:
Inclusion Criteria:

* Meets clinical criteria for Posttraumatic Stress Disorder (PTSD) as per Clinician-Administered PTSD Scale for DSM-5 (CAPS-5)
* TBI present (for PTSD+TBI subjects only) as per American Congress of Rehabilitation Medicine (ACRM) definition
* Mild TBI (for PTSD+TBI subjects only) as per Ohio State University Identification Screener
* Able to provide at least 2 locators
* Able to provide informed consent
* Confirmation that the participant is reliably domiciled
* Agreement to abstain from all other cannabinoid use for the duration of the study
* Willingness to use contraception if of childbearing potential.

Exclusion Criteria:

* History of open head injury
* TBI within the last 6 months
* Moderate or Severe TBI
* SUD in the last 12 months other than mild AUD or nicotine use
* Use of any cannabinoid containing product within the last 1 month
* Positive urine drug screen (Positive for cannabinoids, amphetamine, cocaine, opioids)
* Currently prescribed medications with possible CBD-drug interactions
* Lifetime history of any psychiatric disorder with psychotic features, bipolar disorder
* Exposure to trauma in the last 30 days, including police duty or military service
* Psychotherapy for PTSD or other psychiatric conditions initiated within 2 months of screening
* Not stable for at least 2 months on psychiatric medication, anticonvulsants, antihypertensive medication, sympathomimetic medication, estrogen replacement therapy, medications associated with neurogenesis, or steroid medication
* Active suicide attempt within the past year
* Current significant suicidality (assessed using the C-SSRS), any significant suicidal behavior in the past 12 months, or any history of serious suicide attempts requiring hospitalization, or current significant homicidality.
* Neurologic disorder or systemic illness affecting CNS function (apart from TBI)
* Major medical illness (i.e. cancer or infectious disease.)
* Clinical diagnosis of anemia, advised by physician to avoid blood draws
* Significant laboratory abnormalities, significantly impaired hepatic function, abnormalities in complete blood count or metabolic panel
* Significant allergic reactions to the drug including cannabinoids or sesame oil
* Pregnancy or lactation
* Contraindication to MRI
* Males and females who plan to conceive a child during or two weeks following the study
* Active legal problems likely to result in incarceration within 12 weeks of treatment initiation
* Has a high risk of adverse emotional or behavioral reaction (e.g., evidence of serious personality disorder, antisocial behavior, serious current stressors, and lack of meaningful social support).
* Inpatient psychiatric treatment in past 12 months, with the exception of detox and extended ED stays.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-05-26 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change in PTSD symptoms | Baseline, Week 8
  Baseline - Week 8 change in Clinician-Administered PTSD Scale (CAPS-5) total score. The CAPS-5 is the gold standard clinician administered interview for diagnosing PTSD and assessing symptom severity. Total CAPS-5 scores range from 0-80. Higher scores indicate greater symptom severity.

SECONDARY OUTCOMES:
Change in PTSD symptoms measured with PTSD Checklist (PCL-5) total score. | Weekly over Weeks 1 to 8.
  The PCL-5 is a 20-item self-report measure that assesses DSM-5 symptoms of PTSD. Higher scores indicate greater symptom severity.
Safety and tolerability of cannabidiol | All visits
  Frequency of adverse events collected at all visits following randomization for active arms. The specific tool that will be used to document adverse events is the SAFTEE (Parts A and B).
Change in CAPS-5 symptom cluster severity score for Criterion B, Reexperiencing. | Baseline, Week 8.
  The Criterion B (reexperiencing) severity score is the sum of the individual severity scores for CAPS-5 items 1-5.
Change in CAPS-5 symptom cluster severity score for Criterion C, Avoidance. | Baseline, Week 8.
  The Criterion C (Avoidance) severity score is the sum of the individual severity scores for CAPS-5 items 6 and 7.
Change in CAPS-5 symptom cluster severity score for Criterion D, Negative alterations in cognitions and mood. | Baseline, Week 8.
  The Criterion D (Negative alterations in cognitions and mood) severity score is the sum of the individual severity scores for CAPS-5 items 8-14.
Change in CAPS-5 symptom cluster severity score for Criterion E, Hyperarousal. | Baseline, Week 8.
  The Criterion E (Hyperarousal) severity score is the sum of the individual severity scores for CAPS-5 items 15-20.
Frequency of substantial reduction in PTSD symptoms | Baseline, Week 8
  Number of subjects per arm with a reduction in Baseline - Week 8 CAPS-5 total score equal to or greater than 30%.
Change in plasma CBD levels | Day 1 (post first dose), Week 2, Week 8.
  Peak and trough levels (Cmax) of plasma CBD will be determined via High Performance Liquid Chromatography/Tandem Mass Spectrometry (LC-MS/MS)

CONTACTS AND LOCATIONS:
Overall Officials: Esther M Blessing, MD PhD, Principal Investigator — NYU; Charles R Marmar, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data. Upon reasonable request and to achieve aims in the approved proposal. quests should be directed to Esther.Blessing@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.